CLINICAL TRIAL: NCT04836884
Title: Validation of Core Biopsy of Vascular Anomalies for Clinical Pathology and Genomics
Brief Title: Vascular Anomaly Pathology and Genomics Biopsy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emily C. Bendel, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-011265
Record Dates: First submitted 2021-03-25; First posted 2021-04-08 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Vascular Malformations; Vascular Anomaly; Hemangioma; Arteriovenous Malformations; Venous Malformation; Klippel Trenaunay Syndrome; Lymphatic Malformation
MeSH Terms: conditions — Vascular Malformations; Hemangioma; Arteriovenous Malformations; Klippel-Trenaunay-Weber Syndrome; Lymphatic Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascular anomaly/malformation biopsy (Experimental): Subjects with a vascular anomaly will have a research percutaneous vascular anomaly/malformation biopsy completed at the time of the clinically indicated percutaneous sclerotherapy, embolization and/or ablation.
  Interventions: Procedure: Percutaneous Vascular Anomaly/Malformation Biopsy

INTERVENTIONS:
Procedure: Percutaneous Vascular Anomaly/Malformation Biopsy — US-guided percutaneous vascular anomaly core needle biopsy of up to 10 cores using an 18-gauge co-axial core needle biopsy device at the time of clinically indicated sclerotherapy, embolization or ablation treatment.

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of core biopsy of vascular anomalies for clinical pathology and clinical genomics studies.

DETAILED DESCRIPTION:
Vascular anomalies or vascular malformations often are treated with minimally invasive sclerotherapy, embolization or ablation based on clinical and imaging features without acquisition of tissue. Over the last two decades there have been significant advancements in the understanding of the genetic basis for various vascular anomalies/malformations, which may guide use of therapies for individualized treatment.

As such, given the emergence of novel medications for treatment of vascular anomalies/malformations based on genetic information, acquisition of tissue for pathology and genomic characterization will be increasingly important as treatment of vascular anomalies/vascular malformations moves toward individualized medicine approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and imaging diagnosis of a vascular anomaly.
* No prior treatment for the vascular anomaly.
* Subjects undergoing clinically indicated sclerotherapy, embolization and/or ablation.
* Male or female with age greater than or equal to 18 years.
* Capacity and willingness to provide a written informed consent..

Exclusion Criteria:

* Subjects with prior treatment for their vascular anomaly.
* Uncorrectable coagulopathy.
* Pregnant and/or breast-feeding subjects. A negative pregnancy test within 48 hours of the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Adequacy of core biopsy of vascular anomalies for clinical genomics studies | 18 months
  DNA and RNA will be extracted from the biopsy specimens, undergo qualitative/quantitative quality control assessment and be analyzed by whole genome sequencing (DNA) and RNA sequence analysis (RNA-seq) to determine the adequacy of vascular anomaly biopsy for vascular anomaly genomics characterization.
Adequacy of core biopsy of vascular anomalies for clinical pathology evaluation | 18 months
  Tissue from the vascular anomaly biopsies will undergo histopathology and immunohistochemical staining to determine the adequacy of vascular anomaly core biopsy for clinical pathology characterization.

SECONDARY OUTCOMES:
Safety of vascular anomaly core biopsy | 30 days
  Number of participants with biopsy-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Emily Bendel, MD, Principal Investigator — Mayo Clinic; David A Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials